CLINICAL TRIAL: NCT06390228
Title: Impact of Major Hepatectomy on Recurrence After Resection of Hepatocellular Carcinoma at China Liver Cancer Staging (CNLC) Stage : a Propensity Score Matching Study
Brief Title: Impact of Hepatectomy on HCC Recurrence
Acronym: HCC
Status: Completed | Type: Observational
Sponsor: Anhui Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kunyuan Jiang, Clinical Professor, Anhui Medical University
Other Study IDs: 2023-RE-285; No. 82172071 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma Stage I; Recurrence
Keywords: Hepatocellular Carcinoma; recurrence; hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major hepatectomy: Major hepatectomy was defined as the removal of four or more Couinaud's liver segments.
  Interventions: Procedure: Major hepatectomy
- Minor hepatectomy: Minor hepatectomy was defined as the removal of three or fewer Couinaud's segments.

INTERVENTIONS:
Procedure: Major hepatectomy — the extent of liver resection
  Other Names: minor hepatectomy
  Groups: Major hepatectomy

SUMMARY:
Hepatectomy is the first option for the treatment of hepatocellular carcinoma(HCC) at CNLC Ib stage. HCC patients who undergo curative hepatectomy may experience varying remnant liver volumes and thus leads to different oncological outcomes.

DETAILED DESCRIPTION:
Patients with hepatocellular carcinoma (HCC) who undergo curative hepatectomy may experience varying remnant liver volumes. The investigators aimed to evaluate whether the extent of liver resection has an effect on postoperative recurrence in HCC patients. A retrospective analysis was conducted on 197 patients who underwent hepatectomy for a solitary HCC lesion measuring ≥5 cm between January 2019 and June 2022. Patients were divided into major hepatectomy (MAH) group (n=70) and minor hepatectomy (MIH) group (n=127) based on the extent of liver resection. Recurrence-free survival (RFS) was compared between the two groups. Propensity score matching was employed to mitigate potential biases in this research.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed solitary HCC with a size of ≥5 cm
* Eastern Cooperative Oncology Group score of 0 or 1
* preoperative indocyanine green retention rate at 15 minutes ≤15% and Child-Pugh A classification
* no evidence of vascular invasion or extrahepatic disease.

Exclusion Criteria:

* not diagnosed with HCC or had an HCC measuring <5 cm
* had confirmed tumor metastases or macrovascular invasion based on radiological examinations
* died within 90 days after surgery were excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a final sample of 197 patients was included in this study. Among these patients, 70 underwent MAH (including 62 right hepatectomies, 4 extended right hepatectomies, and 4 extended left hepatectomies), while 127 patients underwent MIH (including 32 left hepatectomies, 10 right anterior hepatectomies, 17 right posterior hepatectomies, 11 mesohepatectomies, 20 left lateral hepatectomies, 21 right partial hepatectomies, 3 left partial hepatectomies, and 13 single segment hepatectomies). Using PSM analysis, 49 pairs of matched patients were identified from each group to compare outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
recurrence-free survival | 2019.1-2023.8
  the time from the time of radical surgery to the time of HCC recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Yin, Ph.D, Study Director — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided